CLINICAL TRIAL: NCT06010173
Title: Efficacy and Safety of Gadopiclenol for Magnetic Resonance Imaging (MRI) in Japanese Adults and Children
Brief Title: Evaluation of Gadopiclenol for Magnetic Resonance Imaging (MRI) in Japanese Adults and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Collaborators: Bracco Imaging S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GDX-44-014 - GDX-101
Record Dates: First submitted 2023-07-28; First posted 2023-08-24 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Lesion in Body Region; CNS Lesion
MeSH Terms: interventions — gadopiclenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adult cohort (Experimental): Each of 2 MRI visits will consist of gadopiclenol injection or comparator injection and MRI procedure (administered in a randomized, blinded and cross-over design). Gadopiclenol and comparator will be injected as a single intravenous (IV) bolus injection at a recommended rate of approximately 2 mL/second followed by a 0.9% saline flush via manual injection or power injector. The injection rate should be identical for both products and may vary depending on scanned organ/region and age of patients.
  Interventions: Drug: Gadopiclenol; Drug: Comparator
- Pediatric cohort (Experimental): Pediatric patients will undergo one MRI examination with gadopiclenol (V2). Gadopiclenol will be injected in a single intravenous (IV) bolus injection at a recommended rate of approximately 2 mL/second followed by a 0.9% saline flush via manual injection or power injector.
  Interventions: Drug: Gadopiclenol
- Pediatric PK cohort (Experimental): Pediatric patients will undergo one MRI examination with gadopiclenol (V2). Gadopiclenol will be injected in a single intravenous (IV) bolus injection at a recommended rate of approximately 2 mL/second followed by a 0.9% saline flush via manual injection or power injector. In addition a total of 3 blood samples per patient will be taken post-injection for PK analysis over the period of 8 hours post-injection.
  Interventions: Drug: Gadopiclenol

INTERVENTIONS:
Drug: Gadopiclenol — Dose/volume of gadopiclenol to be administered will be calculated based on patient's weight at the dose of 0.05 mmol/kg BW
Drug: Comparator — Dose/volume of comparator to be administered will be calculated based on patient's weight at the dose of 0.1 mmol/kg BW
  Arms: Adult cohort

SUMMARY:
This trial conducted in Japan includes 2 different cohorts of patients: adult patients and pediatric patients with two different designs.

* The cohort of adult patients has a prospective, multi-center, randomized, double-blind, controlled, and cross-over design.
* The cohort of pediatric patients has a prospective, multi-center, non-randomized, open-label and single arm design.

Primary objective to demonstrate the non-inferiority of gadopiclenol-enhanced MRI at 0.05 mmol/kg body weight (BW) compared to gadobutrol-enhanced MRI at 0.1 mmol/kg BW in terms of lesion visualization is applicable for adult patients referred for contrast-enhanced MRI of Central Nervous System (CNS) or Body regions.

DETAILED DESCRIPTION:
Adult cohort:

The trial includes a maximum of 5 visits and the record of patient's diagnosis as standard of truth:

* One screening visit (V1) up to 7 days prior to the imaging visit (V2) (V1 can be done on the same day as V2 if all the inclusion/non-inclusion criteria are met).
* Two sequential imaging visits (V2 and V4, minimum interval 2 days and up to 14 days): each visit will consist of gadopiclenol injection or comparator injection and MRI procedure.
* Two safety visits (V3 and V5): 1 day after each injection and MRI examination.

Pediatric cohort:

The inclusions will be divided into 4 age groups: patients from birth to 23 months of age inclusive, patients from 2 to 6 years, patients from 7 to 11 years and patients from 12 to 17 years. The recruitment in the 3 older groups of pediatric patients can be conducted in parallel with adult patients' enrolment. The decision to start the inclusion in the group of patients aged from birth to 23 months will be taken by the Trial Safety Review Board (TSRB).

The trial includes a maximum of 3 visits and the record of patient's diagnosis as standard of truth:

* One screening visit (V1) up to 7 days prior to the imaging visit (V2) (V1 can be done on the same day as V2 if all the inclusion/non-inclusion criteria are met).
* One imaging visit (V2): will consist of gadopiclenol injection and MRI procedure.
* pharmacokinetics (PK) group: Blood sampling for PK will start after gadopiclenol injection according to defined blood sampling schedule and will take up to 8 hours.
* One safety visit (V3): 1 day after gadopiclenol injection and MRI examination.

All Patients:

Images will be assessed off-site in a centralized manner.

Pediatric group :

Up to 24 patients of the pediatric cohort will be included in gadopiclenol PK profile assessment.

The approach implemented for pharmacokinetics (PK) analyses allows sparse blood sampling only and is selected to minimize the clinical burden to children.

All cohorts :

During the trial, the safety of the patients will be monitored and assessed based on the reporting of adverse events (AEs), including vital signs, ECG for pediatric patients and clinical laboratory parameters (blood samples).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for all patients:

  1. All Patient presenting with known or suspected enhancing abnormality(ies) and/or lesion(s) in CNS or in at least one body region among head & neck, thorax (e.g. breast), abdomen (e.g. liver, pancreas and kidney), pelvis (e.g. uterus, ovary and prostate) and musculoskeletal (e.g. extremities) based on a previous imaging procedure performed within 12 months prior to Informed Consent Form (ICF) signature.
  2. All If the patient was treated (either with radiation, surgery, biopsy, or other relevant treatments) between previous imaging evaluation and trial MRI, there should still be a high suspicion of remaining enhancing abnormality(ies) and/or lesion(s) based on available clinical information.
  3. All Patient able and willing to participate in the trial.
  4. All Patient affiliated to national health insurance according to local regulatory requirements.
* Inclusion criteria for adult patients:

  1. A Female or male adult patient having reached legal majority age of 18 years.
  2. A Patient scheduled for a contrast-enhanced MRI examination of CNS or a Body region for clinical reasons and agreeing to have a second contrast-enhanced MRI examination for the purpose of the trial.
  3. A Patient having read the information and having provided his/her consent to participate in writing by dating and signing the informed consent prior to any trial related procedure being conducted.
* Inclusion criteria for pediatric patients:

  1. P Female or male pediatric patient from birth to 17 years. For patients aged from birth to 27 days, only term newborn infants are eligible.

     Patients may not have reached the age of 18 years at the MRI examination.
  2. P Patient whose parent(s) or legal guardian (where applicable) having read the information provided his/her/their consent to patient's participation in writing by dating and signing the informed consent prior to any trial related procedure being conducted.
  3. P Patient with capacity of understanding who received age- and maturity-appropriate information and provided his/her assent to participate in the trial.
  4. P-PK Patient and his/her parent(s) or legal guardian (where applicable) having read the information and provided his/her consent in writing by dating and signing the Informed Consent form or respectively in the patient assent form their consent to participate in the PK analyses.

Exclusion Criteria:

* Non-inclusion criteria for all patients:

  1. bis.All Patient referred for contrast-enhanced cardiac MRI as primary examination (e.g. imaging protocol requiring stress or more than a single injection of gadolinium contrast agent) except for late-enhancement cardiac imaging.

  2.All Patient having received any investigational medicinal product (IMP) within 7 days prior to trial entry or scheduled to receive any investigational treatment during the trial.

  3.All Patient presenting with any contraindication to MRI examinations. 4.All Patient having received any contrast agent (for MRI or CT) within 3 days (or 7 days for patients <1 year old) prior to trial product administration or scheduled to receive any contrast agent during the trial or within 24 hours after the last trial product administration (or 7 days after for patients <1 year old).

  5.All Patient with anticipated, current, or past condition (medical, psychological, social or geographical) that would compromise the patient's safety or her/his ability to participate in the trial in the Investigator's opinion.

  6.All Female patient of childbearing potential with a positive urine pregnancy test done within 1 day prior to each contrast agent administration and not able / not willing to use highly effective birth-controlled method during the trial duration.

Female must have effective medically approved contraception until the last trial visit, if of childbearing potential or with amenorrhea for less than 12 months or must be surgically sterilized or post-menopausal (> 2 years amenorrhea).

7.All Patient unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits and/or unlikelihood of completing the trial.

8.All Patient related to the Investigator or any other trial staff or relative directly involved in the trial conduct.

9.All Patient with known contra-indication(s) to the use or with known sensitivity to one of the products under investigation or to other gadolinium based contrast agents (GBCAs) (such as hypersensitivity, post contrast acute kidney injury).

* Non-inclusion criteria for adult patients:

  1. A Patient with acute disease that may rapidly evolve between the 2 MRI examinations
  2. A Patient previously randomized in this trial.
  3. A Patient expected/scheduled to have any treatment or medical procedure (e.g., chemotherapy, radiotherapy, biopsy, or surgery etc.) that may impact the aspects of the imaged lesions between the 2 MRI examinations. (Patients under corticosteroids and/or maintenance chemotherapy with a stable dose at the time of screening visit and throughout the trial can be included).

  4bis.A Patient presenting an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m^2 (based on Japanese coefficient-modified CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration) formula) assessed within 1 week prior to the first contrast agent administration.
* Non-inclusion criteria for pediatric patients:

  1. P Patient with previously attributed IMP number in this trial.
  2. P Patient with known long QT syndrome.
  3. P Patient presenting an estimated Glomerular Filtration Rate (eGFR) outside age-adjusted normal ranges (based on bedside Schwartz equation) assessed within one week prior to contrast agent administration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Lesion visualization on Paired Images: border delineation | MRI central reading within 2 days to 2 weeks after each MRI exam
  The lesion visualization criterion is based on 3 co-primary criteria rated on a scale from 1 to 4 : border delineation, internal morphology and degree of contrast enhancement assessed by 3 independent off-site blinded readers (IBR).
  The IBR will record each of the 3 co-primary criteria for up to 10 largest and most enhancing lesions on Paired (pre+post) images performed with gadopiclenol and Paired (pre+post) images performed with comparator.
  Delineation of the lesion border is defined as the distinction of lesion from surrounding tissues, structures, or edema, and the detection of extent of the lesion. This criterion will be assessed through the following scale:
  1. = None
  2. = Moderate
  3. = Good
  4. = Excellent
  For each co-primary criterion, a mean of scores will be calculated and will range from 1 to 4.
Lesion visualization on Paired Images: internal morphology | MRI central reading within 2 days to 2 weeks after each MRI exam
  The lesion visualization criterion is based on 3 co-primary criteria rated on a scale from 1 (Poor) to 4 (Excellent): border delineation, internal morphology and degree of contrast enhancement assessed by 3 independent off-site blinded readers (IBR).
  The IBR will record each of the 3 co-primary criteria for up to 10 largest and most enhancing lesions on Paired (pre+post) images performed with gadopiclenol and Paired (pre+post) images performed with comparator.
  Internal morphology of the lesion includes an identification of lesion architecture and the intra-lesion features such as necrosis, hemorrhage, and vascularity. This criterion will be assessed through the following scale:
  1. = Poor
  2. = Moderate
  3. = Good
  4. = Excellent
  For each co-primary criterion, a mean of scores will be calculated and will range from 1 to 4.
Lesion visualization on Paired Images: degree of contrast enhancement | MRI central reading within 2 days to 2 weeks after each MRI exam
  The lesion visualization criterion is based on 3 co-primary criteria rated on a scale from 1 (Poor) to 4 (Excellent): border delineation, internal morphology and degree of contrast enhancement assessed by 3 independent off-site blinded readers (IBR).
  The IBR will record each of the 3 co-primary criteria for up to 10 largest and most enhancing lesions on Paired (pre+post) images performed with gadopiclenol and Paired (pre+post) images performed with comparator.
  This criterion will be a qualitative assessment (not based on signal intensity measurement) according to the following scale:
  1. = No
  2. = Moderate
  3. = Good
  4. = Excellent
  For each co-primary criterion, a mean of scores will be calculated and will range from 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Taoka, MD, Principal Investigator — Nagoya University, JAPAN
Locations (27):
- Japan (27):
  - Shin-Kuki General Hospital, Saitama, Saitama
  - Meitetsu Hospital, Aichi
  - Fukuoka University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Gunma University Hospital, Gunma
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Nakamura Memorial Hospital, Hokkaido
  - National Hospital Organization Shikoku Medical Center for Children and Adults, Kagawa
  - Kanagawa Children's Medical Center, Kanagawa
  - Kobe City Medical Center General Hospital, Kobe
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto City Hospital, Kyoto
  - Tohoku University Hospital, Miyagi
  - Nara Medical University Hospital, Nara
  - Kawasaki Medical School Hospital, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Tominaga Hospital, Osaka
  - Saitama Prefectural Children's Medical Center, Saitama
  - Shizuoka General Hospital, Shizuoka
  - Hamamatsu University Hospital, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - Tokyo Shinagawa Hospital, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - National Center for Child Health and Development, Tokyo
  - Tokyo Metropolitan Children's Medical Center, Tokyo
  - Kurobe City Hospital, Toyama
  - Yamaguchi University Hospital, Yamaguchi

IPD SHARING:
Plan to Share IPD: No